CLINICAL TRIAL: NCT05354466
Title: Effect of Sugammadex Versus Neostigmine on the Occurrence of Respiratory Adverse Events in Children Undergoing Tonsillectomies: a Randomized Controlled Trial
Brief Title: Perioperative Respiratory Adverse events_sugammadex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, Clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2203-061-1305
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Complication
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex as reversal agent (Experimental)
  Interventions: Drug: Sugammadex injection
- Neostigmine as reversal agent (Active Comparator)
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex injection — sugammadex as reversal agent
  Arms: Sugammadex as reversal agent
Drug: Neostigmine — neostigmine as a reversal agent
  Arms: Neostigmine as reversal agent

SUMMARY:
Perioperative respiratory adverse events are common in children. We aimed to evaluate the effect of sugammadex on the incidence of perioperative respiratory adverse events in pediatric patients receiving tonsillectomy

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 2-6 years who were scheduled for tonsillectomy under general anesthesia were enrolled

Exclusion Criteria:

* a recent history of upper respiratory tract infection within 2 weeks of surgery
* allergic reaction to sugammadex
* renal failure
* liver failure
* arrhythmia

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Perioperative respiratory adverse events | from induction of anesthesia to end of operation, about 3 hours
  the incidence of overall perioperative respiratory adverse events; oxygen desaturation < 95%, airway obstruction, laryngospasm, bronchospasm, severe coughing, or postoperative stridor

SECONDARY OUTCOMES:
bradycardia | from induction of anesthesia to end of operation, about 3 hours
  administration of IV atropine, glycopyrrolate, epinephrine, ephedrine
Cardiac arrest | from induction of anesthesia to end of operation, about 3 hours
  documented chest compressions/defibrillation/cardioversion
Anaphylaxis | from induction of anesthesia to end of operation, about 3 hours
  administration of epinephrine, methylprednisolone, diphenhydramine, documented diagnosis of anaphylactic/ anaphylatoid reaction
Allergic reaction | from induction of anesthesia to end of operation, about 3 hours
  redness, urticaria, wheeze
Bronchospasm | from induction of anesthesia to end of operation, about 3 hours
  administration of albuterol, epinephrine
Nausea and vomiting | from induction of anesthesia to end of operation, about 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided